CLINICAL TRIAL: NCT06554769
Title: Efficiency of Rigid Versus Non-rigid Indirect Anchorage During Canine Retraction: A Split Mouth Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed El-Timamy, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo University (CairoU)
Record Dates: First submitted 2024-02-07; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Intervention Model Description: split mouth randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Rigid connection (Experimental): side received a non-rigid 0.014-inch St.St ligature ligating the upper second premolar to the miniscrew.
  Interventions: Procedure: non rigid indirect anchorage connection
- Rigid Connection (Active Comparator): rigid wire 19 x 25 inch stst wire was place between upper first molar and the miniscrew placed between the first molar and second premolar
  Interventions: Procedure: rigid indirect anchorage connection

INTERVENTIONS:
Procedure: non rigid indirect anchorage connection — a nonrigid connection is placed between the miniscrews and the second premolar to prevent mesial tooth movement.
  Arms: Non-Rigid connection
Procedure: rigid indirect anchorage connection — a rigid connection is placed between the miniscrews and the first molar to prevent mesial tooth movement.
  Arms: Rigid Connection

SUMMARY:
Indirect anchorage (In-A) has been broadly used for anchorage reinforcement during anterior segment retraction. The study compared between the efficacy of rigid vs non-rigid connections of In-A i during upper canine retraction in dentoalveolar protrusion cases

DETAILED DESCRIPTION:
Fifteen female patients with dentoalveolar protrusion were included in this study. A miniscrew was inserted following levelling and alignment between the upper first molar and second premolar of both sides. Randomization was applied before first premolar extraction where one side of the arch received a rigid indirect anchorage connection (Group I) of 0.019 x 0.025-inch stainless steel (St.St) archwire from the miniscrew to the auxiliary tube of the upper first molar band, and the other side received a non-rigid indirect anchorage connection (Group II) of 0.014-inch St.St ligature ligating the upper second premolar to the miniscrew. Canine retraction was performed on 0.017 x 0.025-inch St.St archwire applying 1.5 N retraction force. The duration of the study was 7 months. Data was collected from digitized models where anchorage loss of the upper first molar relative to the frontal plane and the vertical position of the upper second premolar were measured

ELIGIBILITY:
Inclusion Criteria:

Adult females Bimaxillary protrusion requiring first premolars extractions Full permanent dentition Good oral hygiene

Exclusion Criteria:

History of previous orthodontic treatment Abnormalities in teeth size and/or shape Vertical, transverse, or anteroposterior skeletal discrepancies Anti-inflammatory medication

Ages: 13 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-02 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
anchorage loss | 4 month
  amount of anchorage loss of the upper first molar during canine retraction using digital model in mm.

SECONDARY OUTCOMES:
vertical position of the upper second premolar | 4 month
  The secondary outcome was to assess the change in the vertical position of the upper second premolar following canine retraction using indirect anchorage using digital models in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt